CLINICAL TRIAL: NCT03908671
Title: Clinical Trial on the Safety and Efficacy of Neoantigen Antigen mRNA Tumor Vaccine in the Treatment of Advanced Esophageal Cancer and Non-small Cell Lung Cancer
Brief Title: Clinical Study of Personalized mRNA Vaccine Encoding Neoantigen in Patients With Advanced Esophageal Cancer and Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stemirna Therapeutics (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STZD-1801
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Cancer; Non Small Cell Lung Cancer
Keywords: mRNA cancer vaccine; cancer vaccine; tumor vaccine; NSCLC; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized mRNA Tumor Vaccine (Experimental): Personalized mRNA Tumor Vaccine Encoding Neoantigen in Patients with advanced esophageal and non-small cell lung cancers
  Interventions: Biological: Personalized mRNA Tumor Vaccine

INTERVENTIONS:
Biological: Personalized mRNA Tumor Vaccine — subcutaneous injection with personalized mRNA tumor vaccine

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety, tolerability and effectiveness of personalized mRNA tumor vaccine encoding neoantigen in Patients with advanced esophageal cancer and non-small cell lung cancer

DETAILED DESCRIPTION:
Primary objectives:

Assessing the safety and tolerability of mRNA personalized tumor vaccines encoding neoantigen for unresectable or metastatic advanced esophageal and non-small cell lung cancers with standard treatment failure or no standard treatment.

Secondary objectives:

Preliminary observation of the efficacy of mRNA personalized tumor vaccines encoding neoantigen for unsurgically resected or metastatic advanced esophageal and non-small cell lung cancers with standard treatment failure or no standard treatment.

Time of tumor progression (TTP); Disease Control Rate (DCR); Objective Remission Rate (ORR); Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 (including both ends), with no gender limit;
* The primary lesion was confirmed by histopathology or cytology as esophageal carcinoma (ⅢC (T4bNanyM0, TanyN3M0), and stage Ⅳ) or non-small cell lung cancer (stage ⅢB-Ⅳ).
* Patients who have metastatic or locally advanced tumor but failed instandard treatments or not suitable for standard treatments;
* According to RECIST (V1.1), the efficacy evaluation criteria for solid tumors, there is at least one measurable lesion.
* Participants with Performance Scale (PS) of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) PS
* Participants must have at least 1 lesion amenable to the mandatory fresh tumor biopsy at study entry
* Fertile patients must agree to use a reliable contraceptive methods (hormonal or barrier methods or abstinence) during the trial and for at least 12 weeks after the last treatment;
* The subject voluntarily participates and signs ICF (Informed consent forms).

Exclusion Criteria:

* Any clinical research drugs, anti-cancer monoclonal antibodies, anti-cancer therapeutic vaccines, immunostimulants (such as IL-2) or using previous investigational drugs within 7 days of the first treatment with mRNA-personalized tumor vaccine or carrelizumab.
* Patients who have allergies or previous history of biological drug allergy;
* Patients who are in pregnant or breast-feeding;
* Patients who are expected to survive less than 3 months during the screening period;
* Tumor mutation load (TMB) is less than 2.0/Mb or tumor neogenic antigen load (TNB) is less than 0.5/Mb or the number of predicted neoantigen is less than 3;
* Patients who underwent major surgery or suffered significant trauma within 4 weeks prior to the enrollment (blood collection), or who are expected to undergo major surgery during the study period;
* Patients with symptoms of brain metastases (Patients with stable brain metastases can be included)
* Extensive lung metastases from tumors, causing breathing difficulties;
* Patients who have tumors close to large blood vessels or nerves;
* A history of severe cardiovascular and cerebrovascular diseases, including but not limited to ventricular arrhythmia requiring clinical intervention; Acute coronary syndrome, myocardial infarction, congestive heart failure, stroke or other grade III and above cardiovascular events within 6 months; New York Heart Association (NYHA) cardiac function grade≥Grade II or left ventricular ejection fraction (LVEF) <50%; Poorly controlled hypertension after standard treatment (systolic blood pressure> 150 mmHg and diastolic blood pressure> 90 mmHg);
* Patients with active ulcers and gastrointestinal bleeding;
* Patients with clinically confirmed autoimmune disease have received systemic treatment in the past 2 years; HIV, HCV positive; HBV-DNA≥1×103 copies/mL (or 2×102 IU/mL); Acute EBV or CMV virus infection;
* Patients with previous history of non-infectious pneumonia requiring steroid therapy or acute lung cancer;
* Participants with a history of interstitial lung disease;
* Patients who have a history of organ transplantation or are waiting for organ transplantation;
* Have any uncontrolled active infection;
* Immunosuppressed subjects, including those with known immunodeficiency; those who are currently using steroids systemically (except those who are using inhaled steroids recently or currently);
* Skin diseases (such as psoriasis) may prevent intradermal vaccines from reaching the target area;
* Who have received chemotherapy, biotherapy, radiotherapy, endocrine therapy, targeted therapy and other tumor treatments, or other experimental drug treatments, or surgery (excluding diagnostic biopsy) within 7 days prior to the first administration of mRNA tumor vaccine treatment;
* Adverse effects from previous antitumor therapy have not recovered referred to CTCAE (V5.0) rating ≤1 (except hair loss);
* The investigator evaluates that the subject is unable or unwilling to comply with the requirements of study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 24 weeks
  During the trial conduction, especially within the 24 weeks of treatment phase when mRNA tumor Vaccine administered, all adverse events (including laboratory abnormality and clinical events) will be closely monitored, and all ≥ grade 3 adverse events per CTCAE will be recorded, including but not limited to the toxicities potentially suspected to relate to injection procedures and/or mRNA Tumor Vaccine therapy as listed below:
  Fever Chills Nausea, vomiting and other gastrointestinal symptoms Fatigue Hypotension Respiratory distress Tumor lysis syndrome Neutropenia, thrombocytopenia Liver and kidney dysfunction Neutropenia, thrombocytopenia Liver and kidney dysfunction

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 1.5 years
  Disease Control Rate of Personalized mRNA Tumor Vaccine
Progression-free Survival (PFS) | 2 years
  Progression-free Survival of Personalized mRNA Tumor Vaccine
Time to Tumor Progression (TTP) | 2 years
  Time to Tumor Progression of Personalized mRNA Tumor Vaccine
Overall Survival (OS) | 3 years
  Overall Survival of Personalized mRNA Tumor Vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided